CLINICAL TRIAL: NCT01066741
Title: Randomized Evaluation of a Phytopharmaceutical in Prevention of Severe Oral Mucositis in Patients Receiving Radiotherapy for Oral Cavity, Oropharynx, Hypopharynx, or Cavum Cancer
Brief Title: Prevention of Radiation-induced Severe Oral Mucositis in Oral Cavity, Oropharynx, Hypopharynx, and Cavum Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: insufficient recruitment, the planed sample size appears not achievable
Sponsor: Centre Leon Berard (Other)
Collaborators: BOIRON (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HOMEODENT; ET2006-042
Record Dates: First submitted 2010-02-05; First posted 2010-02-10 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Oropharynx Cancer; Hypopharynx Cancer
Keywords: Epidermoid carcinoma; Hypopharynx; Oropharynx; Oral cavity; Oral mucosa; Cavum; Severe Oral mucositis; Radiotherapy; Phytotherapy
MeSH Terms: conditions — Oropharyngeal Neoplasms; Hypopharyngeal Neoplasms; Carcinoma, Squamous Cell; Stomatitis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Homeodent® (Experimental): Mouthwash with Homeodent® is started on the first day of irradiation, then continued until the end of the irradiation period or until occurrence of grade ≥3 mucositis. In case of grade ≥3 mucositis, patients are instructed to mouthwash with Sodium Bicarbonate solution until complete disappearance of mucositis or until the end of irradiation.
  Interventions: Drug: Homeodent®
- 1.4 % Sodium Bicarbonate solution (Active Comparator): Mouthwash with sodium bicarbonate is started on the first day of irradiation, then continued until the end of the irradiation period. In case of grade ≥3 mucositis, mouthwash is continued until complete disappearance of the mucositis or until the end of irradiation.
  In both arms, after the end of irradiation, patients can receive treatment with Sodium Bicarbonate solution until complete disappearance of the mucositis.
  Interventions: Drug: 1.4% Sodium Bicarbonate solution

INTERVENTIONS:
Drug: Homeodent® — Two-minute mouthwash with 5 ml of solution diluted in 125 ml of water, 3 times per day after meals and tooth brushing.
  Arms: Homeodent®
Drug: 1.4% Sodium Bicarbonate solution — Two-minute mouthwash with 125 ml of solution, 3 times per day after meals and tooth brushing
  Arms: 1.4 % Sodium Bicarbonate solution

SUMMARY:
The purpose of this study is to evaluate the benefit of a mouthwash with a phytopharmaceutical preparation, Homeodent®, compared to a mouthwash solution containing sodium bicarbonate, for prevention of severe mucositis (grade ≥3, RTOG classification) in patients receiving irradiation for oral cavity, oropharynx, hypopharynx or cavum cancer.

This is a phase III, controlled, randomized, single blind study. The estimated inclusion period is approximately 24 months. The number of patients required in this monocentric study is 330 (165 per arm).

DETAILED DESCRIPTION:
The standard treatment of oral cavity, oropharynx, hypopharynx, and cavum cancers is external radiotherapy. However, one of the associated toxicities is the occurrence of mucositis which can be a limiting factor in the treatment (dose reduction or treatment interruption can limit patient's survival), patient's quality of life decreases and severe complications can occur. The treatment of mucositis is mainly symptomatic; a randomized study has shown a benefit of a mouthwash with Benzydamine, a non steroidal anti-inflammatory drug, for patients receiving 50-Gy radiation. Another study with a lower number of patients has also shown a benefit of using a zinc sulfate solution. Boiron laboratories have developed a phytopharmaceutical preparation, Homeodent®, which has no secondary effects and which could prevent radiation-induced mucositis. This study will evaluate the efficiency of mouthwash with Homeodent® in a large randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient aged ≥ 18 years
* ECOG PS ≤ 2
* Patient with oral cavity and/or oropharynx and/or hypopharynx and/or cavum epidermoid carcinoma, whatever the stage
* Patient receiving a minimum radiation dose of 60 Gy
* Planned radiotherapy to at least 1/3 of the oral mucosa and/or oropharynx
* Mandatory affiliation with a health insurance system
* Signed, written informed consent

Exclusion Criteria:

* Previous irradiation to the oral mucosa and/or oropharynx
* Pre-existing mucositis
* Pregnant or lactating woman (negative serum or urinary pregnancy test for women with child-bearing potential)
* Patient included in another study including experimental radiotherapy possibly toxic to the mucosa
* difficult follow up of the patient
* patient deprived of civil rights

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2009-05; Primary Completion 2011-02 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Rate of occurrence of grade ≥ 3 (RTOG classification) mucositis during irradiation (only the first occurrence will be reported) | At the end of irradiation period (6 weeks)

SECONDARY OUTCOMES:
Rate of grade ≥2 mucositis | At the end of irradiation period (6 weeks)
Rate of Mycosis and Herpes virus infection | At the end of irradiation period (6 weeks)
Rate of use of symptomatic treatment in case of occurrence of mucositis | At the end of irradiation period (6 weeks)
Rate and duration of radiation treatment interruption for toxicity | At the end of irradiation period (6 weeks)
radiation dose, duration of grade ≥3 mucositis, maximum weight loss and maximum level of oral pain in case of grade ≥3 mucositis. | during the occurence of grade≥3 mucositis
Treatment tolerance assessed through a satisfaction questionnaire, and evaluation of compliance | during medication administration
Nutritional intake, estimated using caloric intake and the Detsky score, and rate of enteral and/or parenteral nutrition, in case of toxicity during irradiation | during the period of toxicity
Rate of agreement between the radiation oncologist and the stomatologist for the detection of Grade ≥2 (RTOG classification) mucositis | At the end of irradiation period (6 weeks)
Evaluation of the cost of severe mucositis treatment | during and until the end of severe mucositis treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pascal POMMIER, Principal Investigator — Centre Léon Bérard, Lyon
Locations (1):
- Centre Léon Bérard, Lyon, France

REFERENCES:
- [Background] Trotti A, Bellm LA, Epstein JB, Frame D, Fuchs HJ, Gwede CK, Komaroff E, Nalysnyk L, Zilberberg MD. Mucositis incidence, severity and associated outcomes in patients with head and neck cancer receiving radiotherapy with or without chemotherapy: a systematic literature review. Radiother Oncol. 2003 Mar;66(3):253-62. doi: 10.1016/s0167-8140(02)00404-8. PMID 12742264
- [Background] Scully C, Epstein J, Sonis S. Oral mucositis: a challenging complication of radiotherapy, chemotherapy, and radiochemotherapy: part 1, pathogenesis and prophylaxis of mucositis. Head Neck. 2003 Dec;25(12):1057-70. doi: 10.1002/hed.10318. PMID 14648865
- [Background] Duncan GG, Epstein JB, Tu D, El Sayed S, Bezjak A, Ottaway J, Pater J; National Cancer Institute of Canada Clinical Trials Group. Quality of life, mucositis, and xerostomia from radiotherapy for head and neck cancers: a report from the NCIC CTG HN2 randomized trial of an antimicrobial lozenge to prevent mucositis. Head Neck. 2005 May;27(5):421-8. doi: 10.1002/hed.20162. PMID 15782422
- [Background] Scully C, Epstein J, Sonis S. Oral mucositis: a challenging complication of radiotherapy, chemotherapy, and radiochemotherapy. Part 2: diagnosis and management of mucositis. Head Neck. 2004 Jan;26(1):77-84. doi: 10.1002/hed.10326. PMID 14724910
- [Background] Lapeyre M, Charra-Brunaud C, Kaminsky MC, Geoffrois L, Dolivet G, Toussaint B, Maire F, Pourel N, Simon M, Marchal C, Bey P. [Management of mucositis following radiotherapy for head and neck cancers]. Cancer Radiother. 2001 Nov;5 Suppl 1:121s-130s. French. PMID 11797271
- [Background] Worthington HV, Clarkson JE, Eden OB. Interventions for treating oral mucositis for patients with cancer receiving treatment. Cochrane Database Syst Rev. 2004;(2):CD001973. doi: 10.1002/14651858.CD001973.pub2. PMID 15106165
- [Background] Worthington HV, Clarkson JE, Eden OB. Interventions for preventing oral mucositis for patients with cancer receiving treatment. Cochrane Database Syst Rev. 2006 Apr 19;(2):CD000978. doi: 10.1002/14651858.CD000978.pub2. PMID 16625538
- [Background] Trotti A, Garden A, Warde P, Symonds P, Langer C, Redman R, Pajak TF, Fleming TR, Henke M, Bourhis J, Rosenthal DI, Junor E, Cmelak A, Sheehan F, Pulliam J, Devitt-Risse P, Fuchs H, Chambers M, O'Sullivan B, Ang KK. A multinational, randomized phase III trial of iseganan HCl oral solution for reducing the severity of oral mucositis in patients receiving radiotherapy for head-and-neck malignancy. Int J Radiat Oncol Biol Phys. 2004 Mar 1;58(3):674-81. doi: 10.1016/S0360-3016(03)01627-4. PMID 14967419
- [Background] El-Sayed S, Nabid A, Shelley W, Hay J, Balogh J, Gelinas M, MacKenzie R, Read N, Berthelet E, Lau H, Epstein J, Delvecchio P, Ganguly PK, Wong F, Burns P, Tu D, Pater J. Prophylaxis of radiation-associated mucositis in conventionally treated patients with head and neck cancer: a double-blind, phase III, randomized, controlled trial evaluating the clinical efficacy of an antimicrobial lozenge using a validated mucositis scoring system. J Clin Oncol. 2002 Oct 1;20(19):3956-63. doi: 10.1200/JCO.2002.05.046. PMID 12351592
- [Background] Dodd MJ, Miaskowski C, Greenspan D, MacPhail L, Shih AS, Shiba G, Facione N, Paul SM. Radiation-induced mucositis: a randomized clinical trial of micronized sucralfate versus salt & soda mouthwashes. Cancer Invest. 2003;21(1):21-33. doi: 10.1081/cnv-120016400. PMID 12643006
- [Background] Stokman MA, Spijkervet FK, Burlage FR, Dijkstra PU, Manson WL, de Vries EG, Roodenburg JL. Oral mucositis and selective elimination of oral flora in head and neck cancer patients receiving radiotherapy: a double-blind randomised clinical trial. Br J Cancer. 2003 Apr 7;88(7):1012-6. doi: 10.1038/sj.bjc.6600824. PMID 12671696
- [Background] Saarilahti K, Kajanti M, Joensuu T, Kouri M, Joensuu H. Comparison of granulocyte-macrophage colony-stimulating factor and sucralfate mouthwashes in the prevention of radiation-induced mucositis: a double-blind prospective randomized phase III study. Int J Radiat Oncol Biol Phys. 2002 Oct 1;54(2):479-85. doi: 10.1016/s0360-3016(02)02935-8. PMID 12243825
- [Background] Warde P, O'Sullivan B, Aslanidis J, Kroll B, Lockwood G, Waldron J, Payne D, Bayley A, Ringash J, Kim J, Liu FF, Maxymiw W, Sprague S, Cummings BJ. A Phase III placebo-controlled trial of oral pilocarpine in patients undergoing radiotherapy for head-and-neck cancer. Int J Radiat Oncol Biol Phys. 2002 Sep 1;54(1):9-13. doi: 10.1016/s0360-3016(02)02890-0. PMID 12182969
- [Background] Epstein JB, Silverman S Jr, Paggiarino DA, Crockett S, Schubert MM, Senzer NN, Lockhart PB, Gallagher MJ, Peterson DE, Leveque FG. Benzydamine HCl for prophylaxis of radiation-induced oral mucositis: results from a multicenter, randomized, double-blind, placebo-controlled clinical trial. Cancer. 2001 Aug 15;92(4):875-85. doi: 10.1002/1097-0142(20010815)92:43.0.co;2-1. PMID 11550161
- [Background] Ertekin MV, Koc M, Karslioglu I, Sezen O. Zinc sulfate in the prevention of radiation-induced oropharyngeal mucositis: a prospective, placebo-controlled, randomized study. Int J Radiat Oncol Biol Phys. 2004 Jan 1;58(1):167-74. doi: 10.1016/s0360-3016(03)01562-1. PMID 14697435
- [Background] Maiche AG, Grohn P, Maki-Hokkonen H. Effect of chamomile cream and almond ointment on acute radiation skin reaction. Acta Oncol. 1991;30(3):395-6. doi: 10.3109/02841869109092392. No abstract available. PMID 2036252
- [Background] Fidler P, Loprinzi CL, O'Fallon JR, Leitch JM, Lee JK, Hayes DL, Novotny P, Clemens-Schutjer D, Bartel J, Michalak JC. Prospective evaluation of a chamomile mouthwash for prevention of 5-FU-induced oral mucositis. Cancer. 1996 Feb 1;77(3):522-5. doi: 10.1002/(SICI)1097-0142(19960201)77:33.0.CO;2-6. PMID 8630960